CLINICAL TRIAL: NCT01391507
Title: COR-1, an Anti-Beta1 Receptor Antibody Cyclopeptide in Heart Failure: a Phase II, Multicentre, Randomised, Double-Blind and Placebo-Controlled Study With Parallel Groups
Brief Title: Pilot Study of COR-1 in Heart Failure
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Corimmun GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR100913; 2010-022579-68 (EudraCT Number); COR-1/02
Record Dates: First submitted 2011-07-04; First posted 2011-07-12 (Estimated); Results first posted 2014-08-26 (Estimated); Last update posted 2014-10-17 (Estimated); Status verified 2014-10

CONDITIONS: Cardiomyopathy, Dilated
Keywords: Anti-beta1-receptor autoantibodies; COR-1; Heart failure
MeSH Terms: conditions — Cardiomyopathy, Dilated; Heart Failure | interventions — Sodium Chloride; Standard of Care

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Placebo (Placebo Comparator)
  Interventions: Drug: 0.9 % sodium chloride; Drug: Standard therapy for heart failure
- 20 mg COR-1 (Experimental)
  Interventions: Drug: COR-1; Drug: Standard therapy for heart failure
- 80 mg COR-1 (Experimental)
  Interventions: Drug: COR-1; Drug: Standard therapy for heart failure
- 160 mg COR-1 (Experimental)
  Interventions: Drug: COR-1; Drug: Standard therapy for heart failure

INTERVENTIONS:
Drug: 0.9 % sodium chloride — Monthly intravenous injection for 6 months
  Arms: Placebo
Drug: COR-1 — Monthly intravenous injection for 6 months
  Arms: 160 mg COR-1; 20 mg COR-1; 80 mg COR-1
Drug: Standard therapy for heart failure — All patients will continue to receive standard therapy for heart failure (ie, in accordance with guidelines) throughout the study.

SUMMARY:
The purpose of this study is to investigate the effect of COR-1 in combination with standard therapy in patients with heart failure. The safety and tolerability of COR-1 will also be assessed.

DETAILED DESCRIPTION:
In patients with dilated cardiomyopathy (heart is weakened and enlarged), the presence of anti-beta1-receptor autoantibodies has been shown to predict more depressed left ventricular function, increased prevalence of serious ventricular arrhythmias, sudden cardiac death, and cardiovascular mortality. In animal models, COR-1 cyclopeptide has been shown to bind to, and therefore decrease, the anti-beta1-receptor autoantibody titre. This study will investigate the safety and effectiveness of COR-1 treatment in patients with dilated cardiomyopathy. This study will be a randomized (the study treatment is assigned by chance), double-blind, (neither investigator nor patient knows the treatment that the volunteer receives), multicenter (study is conducted in more than one center) placebo-controlled (one of the treatments is inactive), parallel group study (patients in different treatment groups receive medication at the same time) in men and women who have heart failure due to dilated cardiomyopathy. Eligible patients should also have a left ventricular ejection fraction of less than or equal to 45% (measurement of the percentage of blood leaving the heart each time it contracts) and should be positive for anti-beta1-receptor autoantibodies. The study will consist of 3 phases: a screening phase, a double-blind treatment period, and a follow-up phase. Patients will be randomly assigned to 1 of 4 treatment groups: 20 mg COR-1, 80 mg COR-1, 160 mg COR-1, or placebo (inactive medication). Each patient will receive 1 intravenous dose (medication is injected into a vein) every 4 weeks for a total of 6 months. Patients will come to the study center each time they receive study medication and will remain at the center for 2 to 3 hours following the injection. Blood samples will be drawn at time points during the screening, treatment, and follow-up periods. Patients will return to the study center for follow-up visits at 3 months following completion of the 6-month treatment period. Patients will participate in the study for approximately 9 months. Patient safety will be monitored. The study drug (COR-1) is being investigated for the treatment of heart failure.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed heart failure due to dilated cardiomyopathy with left ventricular ejection fraction < 45%
* Presence of anti-beta1-receptor autoantibodies
* New York Heart Association (NYHA) class II to III heart failure
* Symptomatic heart failure for >1 year and < 8 years
* Treatment with adequate doses of angiotensin converting enzyme inhibitors or angiotensin II receptor blockers, beta-blockers, and optional aldosterone antagonists according to guidelines for at least six months (with the exception of lack of tolerability of any of these drugs) and at stable doses for 2 months prior to screening

Exclusion Criteria:

* Ischemic heart disease characterized by >= 50% coronary artery stenosis and/or history of myocardial infarction
* Third or higher degree valvular defect
* Any disease requiring immunosuppressive drugs (except for <= 5 mg/day prednisone-equivalent dose) or any clinically relevant disorder of the immune system
* History of severe allergies and increased risk for anaphylactic shock (e.g., bronchial asthma)
* History of, or currently active illness, considered to be clinically significant by the Investigator or any other illness that the Investigator considers should exclude the patient from the study or that could interfere with the interpretation of the study results

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2011-10; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Corimmun GmbH Clinical Trial, Study Director — Corimmun GmbH
Locations (4):
- Germany (4):
  - München
  - Regensburg
  - Tübingen
  - Würzburg

REFERENCES:
- [Background] Jahns R, Boivin V, Siegmund C, Inselmann G, Lohse MJ, Boege F. Autoantibodies activating human beta1-adrenergic receptors are associated with reduced cardiac function in chronic heart failure. Circulation. 1999 Feb 9;99(5):649-54. doi: 10.1161/01.cir.99.5.649. PMID 9950662
- [Background] Stork S, Boivin V, Horf R, Hein L, Lohse MJ, Angermann CE, Jahns R. Stimulating autoantibodies directed against the cardiac beta1-adrenergic receptor predict increased mortality in idiopathic cardiomyopathy. Am Heart J. 2006 Oct;152(4):697-704. doi: 10.1016/j.ahj.2006.05.004. PMID 16996841
- [Background] Iwata M, Yoshikawa T, Baba A, Anzai T, Mitamura H, Ogawa S. Autoantibodies against the second extracellular loop of beta1-adrenergic receptors predict ventricular tachycardia and sudden death in patients with idiopathic dilated cardiomyopathy. J Am Coll Cardiol. 2001 Feb;37(2):418-24. doi: 10.1016/s0735-1097(00)01109-8. PMID 11216956
- [Background] Lloyd-Jones D, Adams R, Carnethon M, De Simone G, Ferguson TB, Flegal K, Ford E, Furie K, Go A, Greenlund K, Haase N, Hailpern S, Ho M, Howard V, Kissela B, Kittner S, Lackland D, Lisabeth L, Marelli A, McDermott M, Meigs J, Mozaffarian D, Nichol G, O'Donnell C, Roger V, Rosamond W, Sacco R, Sorlie P, Stafford R, Steinberger J, Thom T, Wasserthiel-Smoller S, Wong N, Wylie-Rosett J, Hong Y; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Heart disease and stroke statistics--2009 update: a report from the American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Circulation. 2009 Jan 27;119(3):480-6. doi: 10.1161/CIRCULATIONAHA.108.191259. No abstract available. PMID 19171871

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Matching placebo (0.9 percent sodium chloride solution) was administered intravenously in addition to the standard therapy for heart failure every 4 weeks for a total of 6 doses.
- COR-1 20 Milligram (mg): COR-1 (JNJ-54452840) was administered at a dose of 20 mg intravenously in addition to the standard therapy for heart failure every 4 weeks for a total of 6 doses.
- COR-1 80 mg: COR-1 was administered at a dose of 80 mg intravenously in addition to the standard therapy for heart failure every 4 weeks for a total of 6 doses.
- COR-1 160 mg: COR-1 was administered at a dose of 160 mg intravenously in addition to the standard therapy for heart failure every 4 weeks for a total of 6 doses.
Period: Overall Study
Arm/Group | Placebo | COR-1 20 Milligram (mg) | COR-1 80 mg | COR-1 160 mg
Started | 10 | 8 | 6 | 12
Completed | 6 | 4 | 2 | 5
Not Completed | 4 | 4 | 4 | 7
Not completed — Death | 0 | 0 | 0 | 1
Not completed — Adverse Event | 1 | 1 | 2 | 2
Not completed — Withdrawal by Subject | 1 | 2 | 1 | 1
Not completed — Lack of Efficacy | 0 | 0 | 0 | 1
Not completed — Protocol Violation | 2 | 1 | 1 | 2

BASELINE CHARACTERISTICS:
Population: Intention-to-treat (ITT) population included all participants who were randomly assigned to treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | COR-1 20 Milligram (mg) | COR-1 80 mg | COR-1 160 mg | Total
Number analyzed (Participants) | 10 | 8 | 6 | 12 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.4 (9.61) | 57.5 (10.92) | 62 (13.59) | 59.8 (11.88) | 59.6 (10.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 1 | 2 | 8
  Male | 7 | 6 | 5 | 10 | 28
Region of Enrollment [Number; unit: participants]
  Germany | 10 | 8 | 6 | 12 | 36

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Left Ventricular Ejection Fraction (LVEF) at Month 6
Description: The LVEF is a fraction of blood (in percent) pumped out of the left ventricle of the heart (the main pumping chamber). Ejection fraction percentages greater than (>) 55% are considered normal. It was measured by biplane echocardiography (central assessment).
Time Frame: Baseline and Month 6
Population: Intention-to-treat (ITT) population included all participants who were randomly assigned to treatment. Missing data was imputed using last observation carried forward (LOCF) method.
Measure: Mean (Standard Deviation); unit: Percentage of blood pumped out
Arm/Group | Placebo | COR-1 20 Milligram (mg) | COR-1 80 mg | COR-1 160 mg
Number analyzed (Participants) | 10 | 8 | 6 | 12
Percentage of blood pumped out
  Baseline | 35.4 (11.72) | 29.4 (12.06) | 35.0 (13.42) | 32.4 (10.77)
  Change at Month 6 | -1.6 (5.94) | 0.8 (5.55) | 5.4 (10.11) | -0.9 (3.09)

2. Secondary Outcome: Change From Baseline in Local Left Ventricular Ejection Fraction (LVEF) at Month 9
Description: The LVEF is a measure of how much blood is pumped out of the left ventricle of the heart (the main pumping chamber). Ejection fraction percentages greater than (>) 55% are considered normal. It was measured by biplane echocardiography (local assessment).
Time Frame: Baseline and Month 9
Population: ITT population included all participants who were randomly assigned to treatment. Missing data was imputed using LOCF method.
Measure: Mean (Standard Deviation); unit: Percentage of blood pumped out
Arm/Group | Placebo | COR-1 20 Milligram (mg) | COR-1 80 mg | COR-1 160 mg
Number analyzed (Participants) | 10 | 8 | 6 | 12
Percentage of blood pumped out
  Baseline | 32.6 (5.78) | 33.6 (9.77) | 35.3 (8.57) | 32.5 (9.27)
  Change at Month 9 | -0.8 (4.39) | -1.9 (5.99) | 3.8 (4.02) | -1.8 (3.13)

3. Secondary Outcome: Change From Baseline in N-Terminal Pro B-Type Natriuretic Peptide (NT-ProBNP) Level at Month 6
Description: The NT-ProBNP is a biomarker (a biologic molecule) that has been shown to predict cardiac events.
Time Frame: Baseline and Month 6
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Picogram (pg)/ Milliliter (mL)
Arm/Group | Placebo | COR-1 20 Milligram (mg) | COR-1 80 mg | COR-1 160 mg
Number analyzed (Participants) | 10 | 8 | 6 | 12
Picogram (pg)/ Milliliter (mL)
  Baseline | 5678.0 (9347.1) | 2215.9 (1692.1) | 971.4 (665.1) | 2299.4 (2024.1)
  Change at Month 6 | -805.7 (1241.0) | 1363.4 (3948.7) | 392.8 (295.7) | 1109.6 (2130.6)

4. Secondary Outcome: Change From Baseline in Central Transmitral Flow Velocity Time Integral (VTI) at Month 6
Description: Transmitral flow VTI measures how blood flows through the heart. This was measured by echocardiogram. Most of the values for transmitral flow VTI were not provided in the reports from central core echocardiographic laboratory due to technical reasons.
Time Frame: Baseline and Month 6
Population: ITT population included all participants who were randomly assigned to treatment. Missing data was imputed using LOCF method. Here, "N" (Number of Participants Analyzed) signifies those participants who were evaluable for this outcome measure. No participants were evaluable for arms COR-1 80 mg and COR-1 160 mg.
Measure: Mean (Standard Deviation); unit: Centimeter (cm)
Arm/Group | Placebo | COR-1 20 Milligram (mg) | COR-1 80 mg | COR-1 160 mg
Number analyzed (Participants) | 2 | 1 | 0 | 0
Centimeter (cm)
  Baseline | 45.0 (31.11) | 21.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. |  |
  Change at Month 6 | 0.0 (0.00) | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. |  |

5. Secondary Outcome: Change From Baseline in Central Tissue E-Wave Doppler Mitral Annular Velocity at Month 6
Description: Tissue doppler mitral annular velocity is a measure of how well the heart fills with blood. This was measured by echocardiogram. Most of the values for E-wave were not provided in the reports from central core echocardiographic laboratory due to technical reasons.
Time Frame: Baseline and Month 6
Population: ITT population included all participants who were randomly assigned to treatment. Missing data was imputed using LOCF method. Here, "N" (Number of Participants Analyzed) signifies those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Centimeter (cm)/ Second (sec)
Arm/Group | Placebo | COR-1 20 Milligram (mg) | COR-1 80 mg | COR-1 160 mg
Number analyzed (Participants) | 5 | 5 | 1 | 4
Centimeter (cm)/ Second (sec)
  Baseline | 5.6 (1.52) | 5.2 (1.10) | 4.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | 5.8 (1.71)
  Change at Month 6 | -0.2 (0.45) | 0.0 (0.00) | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | 0.0 (0.00)

6. Secondary Outcome: Change From Baseline in Distance Walked During Six-minute Walk Test at Month 6
Description: A standardized 6-minute walk test was performed and the distance covered in 6 minutes was measured.
Time Frame: Baseline and Month 6
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Meter
Arm/Group | Placebo | COR-1 20 Milligram (mg) | COR-1 80 mg | COR-1 160 mg
Number analyzed (Participants) | 10 | 8 | 6 | 12
Meter
  Baseline | 421.1 (113.29) | 451.1 (51.02) | 395.2 (81.03) | 420.7 (109.77)
  Change at Month 6 | 38.7 (63.11) | -8.7 (104.35) | 12.8 (57.70) | 2.4 (41.01)

7. Secondary Outcome: Number of Participants With New York Heart Association (NYHA) Classification of Disease Progression
Description: Disease progression (morbidity) was measured by the NYHA classification. The NYHA classification assesses the severity of symptoms of heart failure as judged by the investigator and is comprised of 4 stages. Stage I- No symptoms/limitation in ordinary physical activity (for example, shortness of breath when walking, climbing stairs); Stage II-Mild symptoms (mild shortness of breath and/or angina) and slight limitation during ordinary activity; Stage III- Marked limitation in activity due to symptoms, even during less-than-ordinary activity, (for example, walking short distances [20-100 m]), comfortable only at rest; and Stage IV- Severe limitations in activity/experiences symptoms while at rest (mostly bedbound participants).
Time Frame: Baseline and Month 6
Population: ITT population included all participants who were randomly assigned to treatment. Missing data was imputed using LOCF method. Here 'n' specifies those participants who were evaluated for this outcome measure at given time point.
Measure: Number; unit: Participants
Arm/Group | Placebo | COR-1 20 Milligram (mg) | COR-1 80 mg | COR-1 160 mg
Number analyzed (Participants) | 10 | 8 | 6 | 12
Participants
  Baseline: Stage II (n= 10, 8, 6, 12) | 7 | 8 | 3 | 7
  Baseline: Stage III (n= 10, 8, 6, 12) | 3 | 0 | 3 | 5
  Month 6: Stage I (n= 7, 7, 5, 8) | 1 | 1 | 0 | 0
  Month 6: Stage II (n= 7, 7, 5, 8) | 3 | 4 | 3 | 6
  Month 6: Stage III (n= 7, 7, 5, 8) | 3 | 2 | 2 | 2

8. Secondary Outcome: Change From Baseline in Minnesota Living With Heart Failure Questionnaire Score at Month 6
Description: Minnesota living with heart failure questionnaire is a self-administered, disease-specific measure of health related quality of life (QOL) that assesses participant's perceptions of the influence of heart failure on physical, socioeconomic and psychological aspects of life. Participants responded to 21 items using a six-point response scale (0-5). The total summary score can range from 0-105 with a lower score reflecting better heart failure related QOL.
Time Frame: Baseline and Month 6
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | COR-1 20 Milligram (mg) | COR-1 80 mg | COR-1 160 mg
Number analyzed (Participants) | 7 | 7 | 5 | 11
Units on a scale
  Baseline | 23.7 (11.57) | 21.4 (12.09) | 33.2 (23.09) | 25.9 (25.27)
  Change at Month 6 | 3.3 (10.70) | 3.3 (16.25) | 1.8 (9.50) | 2.4 (20.50)

9. Secondary Outcome: Change From Baseline in Holter Electrocardiography (ECG) Parameters (Heart Rate) at Month 6
Description: A Holter monitor is a portable device which monitors the electrical activity (electrocardiography) of the heart. Mean heart rate, maximum heart rate and minimum heart rate were evaluated.
Time Frame: Baseline and Month 6
Population: Safety population included all participants who received at least 1 dose of the study agent.
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Placebo | COR-1 20 Milligram (mg) | COR-1 80 mg | COR-1 160 mg
Number analyzed (Participants) | 7 | 7 | 5 | 11
Beats per minute
  Baseline: Mean Heart Rate | 74.6 (7.00) | 76.9 (10.92) | 84.2 (11.43) | 75.3 (8.59)
  Change at Month 6: Mean Heart Rate | 1.3 (6.68) | -0.9 (3.63) | -5.8 (10.18) | 1.4 (6.97)
  Baseline: Maximum Heart Rate | 126.4 (18.28) | 130.3 (33.26) | 123.0 (15.26) | 125.1 (35.23)
  Change at Month 6: Maximum Heart Rate | -0.8 (15.24) | 5.4 (40.15) | 0.0 (25.30) | -2.0 (31.56)
  Baseline: Minimum Heart Rate | 51.6 (11.54) | 59.3 (13.12) | 66.0 (4.16) | 58.7 (6.65)
  Change at Month 6: Minimum Heart Rate | 0.5 (3.39) | 0.1 (3.93) | -7.8 (4.50) | -2.3 (10.09)

10. Secondary Outcome: Number of Participants With Holter Electrocardiography (ECG) Parameters
Description: A Holter monitor is a portable device which monitors the electrical activity (electrocardiography) of the heart. Block, Heart rhythm, AV junctional, Ventricular, Lown classification, Results were evaluated.
Time Frame: Baseline and Month 6
Population: Safety population included all participants who received at least 1 dose of the study agent.
Measure: Number; unit: Participants
Arm/Group | Placebo | COR-1 20 Milligram (mg) | COR-1 80 mg | COR-1 160 mg
Number analyzed (Participants) | 7 | 7 | 5 | 11
Participants
  Baseline: No block | 7 | 7 | 5 | 7
  Baseline: AV block I | 0 | 0 | 0 | 3
  Baseline: AV block II | 0 | 0 | 0 | 0
  Baseline: AV block III | 0 | 0 | 0 | 0
  Baseline: Sinus rhythm | 5 | 4 | 4 | 7
  Baseline: Atrial fibrillation | 0 | 0 | 0 | 0
  Baseline:Atrial fibrillation-paroxysmal/persistent | 2 | 1 | 1 | 1
  Baseline: Other | 0 | 2 | 0 | 2
  Baseline; AV junctional, 0-240/24h | 5 | 6 | 4 | 6
  Baseline: AV junctional, 241-1000/24h | 2 | 0 | 0 | 3
  Baseline: AV junctional, 1001-2400/24h | 0 | 0 | 1 | 1
  Baseline: Ventricular, 0-240/24h | 1 | 1 | 1 | 4
  Baseline: Ventricular, 241-1000/24h | 2 | 2 | 2 | 1
  Baseline: Ventricular, 1001-2400/24h | 4 | 3 | 2 | 5
  Baseline: 0 No VES | 0 | 1 | 0 | 0
  Baseline: I Occasional individual VES (< 30/h) | 3 | 0 | 1 | 4
  Baseline: II Frequent VES (>30/h) | 0 | 2 | 0 | 0
  Baseline: IIIa Polymorphous VES | 1 | 0 | 0 | 1
  Baseline: IIIb Ventricular bigeminy | 0 | 0 | 0 | 1
  Baseline: IVa Couplets, repetitive VES | 1 | 2 | 2 | 1
  Baseline: IVb Runs, repetitive VES | 2 | 2 | 1 | 3
  Baseline: V Early occurring VES(R-on T phenomenon) | 0 | 0 | 0 | 0
  Baseline: II, IIIa, IVa, IVb | 0 | 0 | 1 | 0
  Baseline: Normal | 2 | 0 | 2 | 1
  Baseline: Abnormal, NCS | 5 | 5 | 1 | 8
  Baseline: Abnormal, CS | 0 | 2 | 2 | 1
  Month 6: No block | 6 | 7 | 5 | 5
  Month 6: AV block I | 0 | 0 | 0 | 1
  Month 6: AV block II | 0 | 0 | 0 | 1
  Month 6: AV block III | 0 | 0 | 0 | 0
  Month 6: Sinus rhythm | 2 | 4 | 3 | 6
  Month 6: Atrial fibrillation | 0 | 0 | 0 | 0
  Month 6: Atrial fibrillation-paroxysmal/persistent | 2 | 2 | 1 | 0
  Month 6: Other | 2 | 1 | 1 | 1
  Month 6: AV junctional, 0-240/24h | 5 | 5 | 4 | 4
  Month 6: AV junctional, 241-1000/24h | 1 | 2 | 1 | 1
  Month 6: AV junctional, 1001-2400/24h | 0 | 0 | 0 | 2
  Month 6: Ventricular, 0-240/24h | 2 | 2 | 1 | 2
  Month 6: Ventricular, 241-1000/24h | 0 | 2 | 1 | 1
  Month 6: Ventricular, 1001-2400/24h | 4 | 3 | 3 | 4
  Month 6: 0 No VES | 0 | 1 | 0 | 0
  Month 6: I Occasional individual VES (< 30/h) | 2 | 0 | 2 | 2
  Month 6: II Frequent VES (>30/h) | 0 | 0 | 0 | 1
  Month 6: IIIa Polymorphous VES | 2 | 3 | 1 | 1
  Month 6: IVa Couplets, repetitive VES | 1 | 1 | 0 | 1
  Month 6: IVb Runs, repetitive VES | 1 | 1 | 1 | 2
  Month 6: V Early occurring VES (R-on T phenomenon) | 0 | 0 | 0 | 0
  Month 6: II, IIIa, IVa, IVb | 0 | 1 | 1 | 0
  Month 6: Normal | 0 | 0 | 1 | 1
  Month 6: Abnormal, NCS | 6 | 6 | 3 | 5
  Month 6: Abnormal, CS | 0 | 1 | 1 | 1

ADVERSE EVENTS:
Time Frame: 9 months
Arm/Group | Placebo | COR-1 20 Milligram (mg) | COR-1 80 mg | COR-1 160 mg
Serious Adverse Events (participants affected / at risk) | 1/10 | 1/8 | 1/6 | 6/12
Other Adverse Events (participants affected / at risk) | 4/10 | 7/8 | 5/6 | 6/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=10) | COR-1 20 Milligram (mg) (N=8) | COR-1 80 mg (N=6) | COR-1 160 mg (N=12)
Cardiac Failure (Cardiac disorders) | 1 | 0 | 1 | 2
Cardiogenic Shock (Cardiac disorders) | 0 | 0 | 0 | 1
Heart Valve Incompetence (Cardiac disorders) | 0 | 0 | 0 | 1
Sinus Arrest (Cardiac disorders) | 0 | 0 | 0 | 1
Cardiac Death (General disorders) | 0 | 0 | 0 | 1
Lobar Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1
Ejection Fraction Decreased (Investigations) | 0 | 0 | 0 | 1
Weight Increased (Investigations) | 1 | 0 | 0 | 0
Ovarian Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Loss of Consciousness (Nervous system disorders) | 0 | 0 | 0 | 1
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 1
Mental Disorder (Psychiatric disorders) | 0 | 0 | 0 | 1
Renal Failure (Renal and urinary disorders) | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Haemodialysis (Surgical and medical procedures) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=10) | COR-1 20 Milligram (mg) (N=8) | COR-1 80 mg (N=6) | COR-1 160 mg (N=12)
Arrhythmia (Cardiac disorders) | 0 | 1 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 1 | 0 | 0
Cardiac Failure (Cardiac disorders) | 1 | 1 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 1 | 0 | 0
Sinus Bradycardia (Cardiac disorders) | 0 | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0
Ventricular Extrasystoles (Cardiac disorders) | 0 | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Abdominal Pain Lower (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Abdominal Pain Upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Anal Inflammation (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Nausea (Gastrointestinal disorders) | 1 | 1 | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 1
Chest Pain (General disorders) | 0 | 0 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 0 | 1
General Physical Health Deterioration (General disorders) | 0 | 0 | 0 | 1
Injection Site Haematoma (General disorders) | 1 | 0 | 0 | 0
Oedema Peripheral (General disorders) | 1 | 0 | 2 | 0
Pyrexia (General disorders) | 1 | 0 | 1 | 1
Hepatomegaly (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Acute Tonsillitis (Infections and infestations) | 1 | 0 | 0 | 0
Cystitis (Infections and infestations) | 1 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 1 | 2 | 1
Oral Herpes (Infections and infestations) | 0 | 1 | 0 | 0
Respiratory Tract Infection (Infections and infestations) | 1 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 1 | 1
Staphylococcal Infection (Infections and infestations) | 0 | 0 | 1 | 0
Excoriation (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Face Injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Traumatic Haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Blood Creatine Increased (Investigations) | 0 | 1 | 0 | 0
Blood Potassium Increased (Investigations) | 0 | 1 | 0 | 1
Blood Pressure Decreased (Investigations) | 0 | 1 | 0 | 0
Carotid Bruit (Investigations) | 0 | 0 | 1 | 0
Glomerular Filtration Rate Abnormal (Investigations) | 0 | 0 | 1 | 0
Heart Rate Increased (Investigations) | 1 | 1 | 1 | 1
Hepatic Enzyme Increased (Investigations) | 0 | 0 | 1 | 0
Prostatic Specific Antigen Increased (Investigations) | 0 | 0 | 0 | 1
Weight Increased (Investigations) | 1 | 0 | 0 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Gout (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Joint Swelling (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Aura (Nervous system disorders) | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 1 | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 1
Presyncope (Nervous system disorders) | 0 | 0 | 1 | 0
Sciatica (Nervous system disorders) | 1 | 0 | 0 | 1
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0
Hallucination (Psychiatric disorders) | 0 | 0 | 0 | 1
Mental Disorder (Psychiatric disorders) | 0 | 0 | 0 | 1
Renal Impairment (Renal and urinary disorders) | 1 | 0 | 1 | 0
Gynaecomastia (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 2
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Wisdom Teeth Removal (Surgical and medical procedures) | 0 | 0 | 0 | 1
Venous Insufficiency (Vascular disorders) | 1 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
Due to the decision to amend protocol to a pilot study coupled with the high study agent discontinuation rate, safety or efficacy of JNJ-54452840 could not be concluded due to the insufficient sample size and drug exposure to investigational agent.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If Sponsor should have justified objections, then Hospital will respond to these objections as the scientific nature of publication are not negatively affected. If no agreement can be reached, they will appeal to an independent body of experts to resolve the points in dispute. It is not permissible to publish study data before overall study results are published without the written consent of Sponsor. However, this applies to a maximum period of 12 months after study has ended or been cancelled.